CLINICAL TRIAL: NCT02974153
Title: A Parallel Group, Double-Blind, Randomized, Placebo Controlled Phase 3 Trial to Evaluate the Efficacy and Safety of ALD403 Administered Intravenously in Patients With Chronic Migraine
Brief Title: Evaluation of ALD403 (Eptinezumab) in the Prevention of Chronic Migraine
Acronym: PROMISE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alder Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ALD403-CLIN-011
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ALD403 (Eptinezumab) Dose Level 1 (Experimental): ALD403 (Eptinezumab) Dose Level 1 (IV)
  Interventions: Biological: ALD403 (Eptinezumab)
- ALD403 (Eptinezumab) Dose Level 2 (Experimental): ALD403 (Eptinezumab) Dose Level 2 (IV)
  Interventions: Biological: ALD403 (Eptinezumab)
- Placebo (Placebo Comparator): Placebo (IV)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ALD403 (Eptinezumab)
  Other Names: Eptinezumab-jjmr; Vyepti
  Arms: ALD403 (Eptinezumab) Dose Level 1; ALD403 (Eptinezumab) Dose Level 2
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of ALD403 in the prevention of migraine headache in chronic migraineurs.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age, inclusive, who were diagnosed with migraines at ≤ 50 years of age, and have a history of chronic migraine for ≥ 12 months before screening.
* During the 28 day screening period, subjects must adequately complete the headache eDiary and must have headaches occurring on ≥ 15 to ≤ 26 days of which at least 8 must be migraine days.
* Headache eDiary was completed on at least 24 of the 28 days prior to randomization.

Exclusion Criteria:

* Confounding and clinically significant pain syndromes (e.g. fibromyalgia, chronic low back pain, complex regional pain syndrome).
* Psychiatric conditions that are uncontrolled and/or untreated, including conditions that are not controlled for a minimum of 6 months prior to screening. Patients with a lifetime history of psychosis, mania, or dementia are excluded.
* Any use of botulinum toxin for migraine or for any other medical/cosmetic reasons requiring injections within 4 months prior to screening and during the screening period.
* History or diagnosis of complicated migraine (ICHD-III beta version, 20134), chronic tension-type headache, hypnic headache, cluster headache, hemicrania continua, new daily persistent headache, or sporadic and familial hemiplegic migraine.
* Receipt of any monoclonal antibody treatment (within or outside a clinical trial) within 6 months before screening.
* Previously dosed with ALD403 or any monoclonal antibody targeting the CGRP pathway.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1121 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (124):
- United States (68):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Carlsbad, California
  - Research Site, Oceanside, California
  - Research Site, Orange, California
  - Research Site, Oxnard, California
  - Research Site, Palo Alto, California
  - Research Site, Redlands, California
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Torrance, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, New London, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Overland Park, Kansas
  - Research Site, Prairie Village, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Marrero, Louisiana
  - Research Site, Waldorf, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, North Attleboro, Massachusetts
  - Research Site, Watertown, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Flowood, Mississippi
  - Research Site, City of Saint Peters, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Lebanon, New Hampshire
  - Research Site, Princeton, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Amherst, New York
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Plainview, New York
  - Research Site, Rochester, New York
  - Research Site, Durham, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Scottdale, Pennsylvania
  - Research Site, Smithfield, Pennsylvania
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Richmond, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Spokane, Washington
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Liège
- Czechia (3):
  - Research Site, Brno
  - Research Site, Choceň
  - Research Site, Prague
- Denmark (2):
  - Research Site, Glostrup Municipality
  - Research Site, Viborg
- Research Site, Tbilisi, Georgia
- Germany (5):
  - Research Site, Berlin
  - Research Site, Erlangen
  - Research Site, Hamburg
  - Research Site, Nordheim
  - Research Site, Unterhaching
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Pécs
- Italy (5):
  - Research Site, Ancona
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Pavia
  - Research Site, Roma
- Russia (7):
  - Research Site, Kazan'
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Slovakia (4):
  - Research Site, Banská Bystrica
  - Research Site, Dolný Kubín
  - Research Site, Dubnica nad Váhom
  - Research Site, Krompachy
- Spain (11):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Guadalajara
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Navarrés
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Terrassa
  - Research Site, Valencia
  - Research Site, Valladolid
- Ukraine (8):
  - Research Site, Dnipro
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya
- United Kingdom (6):
  - Research Site, Glasgow
  - Research Site, Inverness
  - Research Site, London
  - Research Site, Newcastle
  - Research Site, Salford
  - Research Site, Stoke-on-Trent

REFERENCES:
- [Derived] Tepper SJ, Diamond ML, Hirman J, Asher D, Fiore D, Cady R. Eptinezumab treatment was associated with longer interictal headache/migraine periods which corresponded to greater improvements in patient-reported quality of life measures. J Neurol. 2024 Dec 12;272(1):4. doi: 10.1007/s00415-024-12809-z. PMID 39666143
- [Derived] Kaniecki RG, Friedman DI, Asher D, Hirman J, Cady R. Improving to Four or Fewer Monthly Headache Days Per Month Provides a Clinically Meaningful Therapeutic Target for Patients with Chronic Migraine. Pain Ther. 2023 Oct;12(5):1179-1194. doi: 10.1007/s40122-023-00525-x. Epub 2023 Jun 28. PMID 37378754
- [Derived] Pozo-Rosich P, Dodick DW, Ettrup A, Hirman J, Cady R. Shift in diagnostic classification of migraine after initiation of preventive treatment with eptinezumab: post hoc analysis of the PROMISE studies. BMC Neurol. 2022 Oct 25;22(1):394. doi: 10.1186/s12883-022-02914-9. PMID 36284281
- [Derived] Cowan RP, Marmura MJ, Diener HC, Starling AJ, Schim J, Hirman J, Brevig T, Cady R. Quantity changes in acute headache medication use among patients with chronic migraine treated with eptinezumab: subanalysis of the PROMISE-2 study. J Headache Pain. 2022 Sep 6;23(1):115. doi: 10.1186/s10194-022-01482-0. PMID 36068494
- [Derived] Apelian R, Boyle L, Hirman J, Asher D. Measuring dose-related efficacy of eptinezumab for migraine prevention: post hoc analysis of PROMISE-1 and PROMISE-2. J Headache Pain. 2022 Apr 18;23(1):48. doi: 10.1186/s10194-022-01418-8. PMID 35436857
- [Derived] McAllister P, Kudrow D, Cady R, Hirman J, Ettrup A. Reduction in migraine-associated burden after eptinezumab treatment in patients with chronic migraine. Cephalalgia. 2022 Sep;42(10):1005-1012. doi: 10.1177/03331024221089567. Epub 2022 Mar 25. PMID 35332807
- [Derived] Ashina M, McAllister P, Cady R, Hirman J, Ettrup A. Efficacy and safety of eptinezumab in patients with migraine and self-reported aura: Post hoc analysis of PROMISE-1 and PROMISE-2. Cephalalgia. 2022 Jul;42(8):696-704. doi: 10.1177/03331024221077646. Epub 2022 Mar 18. PMID 35302389
- [Derived] Buse DC, Winner PK, Charleston L 4th, Hirman J, Cady R, Brevig T. Early response to eptinezumab indicates high likelihood of continued response in patients with chronic migraine. J Headache Pain. 2022 Feb 21;23(1):29. doi: 10.1186/s10194-022-01387-y. PMID 35189811
- [Derived] Martin V, Nagy AJ, Janelidze M, Giorgadze G, Hirman J, Cady R, Mehta L, Buse DC. Impact of Baseline Characteristics on the Efficacy and Safety of Eptinezumab in Patients With Migraine: Subgroup Analyses of PROMISE-1 and PROMISE-2. Clin Ther. 2022 Mar;44(3):389-402. doi: 10.1016/j.clinthera.2022.01.006. Epub 2022 Feb 5. PMID 35131090
- [Derived] Lipton RB, Charleston L 4th, Tassorelli C, Brevig T, Hirman J, Cady R. Patient-reported outcomes, health-related quality of life, and acute medication use in patients with a >/= 75% response to eptinezumab: subgroup pooled analysis of the PROMISE trials. J Headache Pain. 2022 Feb 7;23(1):23. doi: 10.1186/s10194-022-01386-z. PMID 35130836
- [Derived] Smith TR, Spierings ELH, Cady R, Hirman J, Ettrup A, Shen V. Cardiovascular outcomes in adults with migraine treated with eptinezumab for migraine prevention: pooled data from four randomized, double-blind, placebo-controlled studies. J Headache Pain. 2021 Nov 25;22(1):143. doi: 10.1186/s10194-021-01360-1. PMID 34823467
- [Derived] Smith TR, Spierings ELH, Cady R, Hirman J, Schaeffler B, Shen V, Sperling B, Brevig T, Josiassen MK, Brunner E, Honeywell L, Mehta L. Safety and tolerability of eptinezumab in patients with migraine: a pooled analysis of 5 clinical trials. J Headache Pain. 2021 Mar 30;22(1):16. doi: 10.1186/s10194-021-01227-5. PMID 33781209
- [Derived] Silberstein S, Diamond M, Hindiyeh NA, Biondi DM, Cady R, Hirman J, Allan B, Pederson S, Schaeffler B, Smith J. Eptinezumab for the prevention of chronic migraine: efficacy and safety through 24 weeks of treatment in the phase 3 PROMISE-2 (Prevention of migraine via intravenous ALD403 safety and efficacy-2) study. J Headache Pain. 2020 Oct 6;21(1):120. doi: 10.1186/s10194-020-01186-3. PMID 33023473
- [Derived] Lipton RB, Goadsby PJ, Smith J, Schaeffler BA, Biondi DM, Hirman J, Pederson S, Allan B, Cady R. Efficacy and safety of eptinezumab in patients with chronic migraine: PROMISE-2. Neurology. 2020 Mar 31;94(13):e1365-e1377. doi: 10.1212/WNL.0000000000009169. Epub 2020 Mar 24. PMID 32209650

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2263 participants signed the ICF, of which 1121 participants met the entry criteria and were randomized into the trial.
Groups:
- 300 mg ALD403: Participants were randomized to receive a single 300 mg IV infusion of ALD403 on Days 0 and 84 (Week 12).
- 100 mg ALD403: Participants were randomized to receive a single 100 mg IV infusion of ALD403 on Days 0 and 84 (Week 12).
- Placebo: Participants were randomized to receive a single placebo IV infusion on Days 0 and 84 (Week 12).
Period: Overall Study
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Started | 374 | 372 | 375
Participants Treated | 350 | 356 | 366
Completed | 322 | 324 | 325
Not Completed | 52 | 48 | 50
Not completed — Adverse Event | 6 | 0 | 1
Not completed — Lack of Efficacy | 6 | 5 | 10
Not completed — Lost to Follow-up | 9 | 10 | 17
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Withdrawal by Subject | 9 | 16 | 11
Not completed — Study Burden | 8 | 7 | 3
Not completed — Other | 14 | 8 | 7

BASELINE CHARACTERISTICS:
Population: Safety population includes all participants who received study drug or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo | Total
Number analyzed (Participants) | 350 | 356 | 366 | 1072
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (10.36) | 41.0 (11.72) | 39.6 (11.28) | 40.5 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314 | 307 | 325 | 946
  Male | 36 | 49 | 41 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 33 | 35 | 86
  Not Hispanic or Latino | 332 | 323 | 331 | 986
  Unknown or Not Reported | 0 | 00 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 23 | 21 | 38 | 82
  White | 322 | 332 | 321 | 975
  More than one race | 2 | 1 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Hungary | 3 | 5 | 3 | 11
  United States | 195 | 198 | 232 | 625
  Czechia | 12 | 7 | 8 | 27
  Ukraine | 34 | 43 | 33 | 110
  United Kingdom | 3 | 4 | 2 | 9
  Spain | 18 | 22 | 18 | 58
  Russia | 32 | 27 | 27 | 86
  Belgium | 0 | 0 | 1 | 1
  Denmark | 3 | 2 | 1 | 6
  Italy | 7 | 3 | 5 | 15
  Georgia | 36 | 38 | 23 | 97
  Slovakia | 4 | 5 | 8 | 17
  Germany | 3 | 2 | 5 | 10
Baseline Migraine Days [Count of Participants; unit: Participants]
  Less than 17 days per month | 197 | 199 | 206 | 602
  Greater than or equal to 17 days per month | 153 | 157 | 160 | 470
Medication overuse headache diagnosis [Count of Participants; unit: Participants]
  No | 203 | 217 | 221 | 641
  Yes | 147 | 139 | 145 | 431

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Monthly Migraine Days
Description: Monthly migraine days are summarized in 28-day intervals, and averaged across Weeks 1-12
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Full Range); unit: Migraine Days
Groups:
- 300 mg ALD403: Participants received a single 300 mg IV infusion of ALD403 on Days 0 and 84 (Week 12).
- 100 mg ALD403: Participants received a single 100 mg IV infusion of ALD403 on Days 0 and 84 (Week 12).
- Placebo: Participants received a single placebo IV infusion on Days 0 and 84 (Week 12).
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
Migraine Days | -8.2 [-23 to 11] | -7.7 [-22 to 10] | -5.6 [-25 to 9]
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -2.60, 95% CI 2-sided [-3.45 to -1.74], Standard Deviation 6.15
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -2.03, 95% CI 2-sided [-2.88 to -1.18], Standard Deviation 6.15

2. Secondary Outcome: 75% Migraine Responder Rate
Description: Participants with an average reduction in migraine days of at least 75% over Weeks 1 to 12, as compared with baseline.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
Participants | 116 | 95 | 55
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 18.1, 95% CI 2-sided [12.0 to 24.3]
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 11.7, 95% CI 2-sided [5.8 to 17.5]

3. Secondary Outcome: 75% Migraine Responder Rate - 4 Week
Description: Participants with an average reduction in migraine days of at least 75% over Weeks 1 to 4, as compared with baseline.
Time Frame: Week 1-4
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
Participants | 129 | 110 | 57
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 21.3, 95% CI 2-sided [15.0 to 27.6]
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.3, 95% CI 2-sided [9.3 to 21.4]

4. Secondary Outcome: 50% Migraine Responder Rate
Description: Participants with an average reduction in migraine days of at least 50% over Weeks 1 to 12, as compared with baseline.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
Participants | 215 | 205 | 144
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 22.1, 95% CI 2-sided [14.9 to 29.2]
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 18.2, 95% CI 2-sided [11.1 to 25.4]

5. Secondary Outcome: Percentage of Participants With a Migraine on the Day After Dosing
Description: The percentage of participants with a migraine on the day after dosing, where Day 0 is treatment Day and Day 1 is the day after dosing.
Time Frame: Day 1
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Number; unit: Percentage of participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
Percentage of participants | 27.8 | 28.6 | 42.3
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Change in Monthly Acute Medication Days
Description: An acute medication migraine day was a day with any triptan or ergotamine use as recorded in the eDiary.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: Acute Medication Migraine Days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
Acute Medication Migraine Days | -3.5 (4.62) | -3.3 (4.89) | -1.9 (4.18)
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-1.88 to -0.87]
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-1.66 to -0.65]

7. Secondary Outcome: Change From Baseline of Headache Impact Test (HIT-6) Score
Description: The HIT-6 measures the impact of headache on the participant's functional health and well-being in 6 domains: pain; role functioning (ability to carry out usual activities); social functioning; energy or fatigue; cognition; and emotional distress assessed over the prior 12-week period. The total possible scores range from 36 (no impact) to 78 (worst impact).
Time Frame: Baseline to Week 12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
score on a scale | -7.3 [-40 to 10] | -6.2 [-34 to 10] | -4.5 [-32 to 15]
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -2.88, 95% CI 2-sided [-3.91 to -1.84]
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p = 0.0010, ANCOVA; Mean Difference (Final Values) = -1.73, 95% CI 2-sided [-2.76 to -0.70]

8. Secondary Outcome: Change in Migraine Prevalence From Baseline to Week 4
Description: The avarage change in percentage of participants with a migraine on any given day during baseline and the equivalent avarage rate over Weeks 1-4.
Time Frame: Baseline to Week 4
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (95% Confidence Interval); unit: percentage of participants with migraine
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
percentage of participants with migraine | -29.8 [-32.10 to -27.49] | -27.1 [-29.35 to -24.78] | -18.8 [-21.06 to -16.54]
Statistical Analysis 1: Comparison: 300 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, Repeated Measures Model; Mean Difference (Final Values) = -11.00, 95% CI 2-sided [-14.22 to -7.77]
Statistical Analysis 2: Comparison: 100 mg ALD403 vs Placebo; Test type: Superiority; p < 0.0001, Repeated Measures Model; Mean Difference (Final Values) = -8.26, 95% CI 2-sided [-11.48 to -5.05]

9. Secondary Outcome: 75% Headache Responder Rate
Description: Participants with an average reduction in headache days of at least 75% over Weeks 1 to 12, as compared with baseline.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
Participants | 61 | 49 | 29

10. Secondary Outcome: 50% Headache Responder Rate
Description: Participants with an average reduction in headache days of at least 50% over Weeks 1 to 12, as compared with baseline.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
Participants | 169 | 150 | 95

11. Secondary Outcome: 100% Migraine Responder Rate
Description: For each 4-week period the 100% response is determined, and the result for a participant is the average rate across Weeks 1-12. If a participant has one 4-week period out of 3 with 100% response, they are included as 33%.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Number; unit: percent of participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
percent of participants | 15.1 | 10.8 | 5.1

12. Secondary Outcome: 100% Headache Responder Rate
Description: as for outcome 11
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Number; unit: Percent of participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
Percent of participants | 3.8 | 2.0 | 1.5

13. Secondary Outcome: Change From Baseline in Monthly Migraine Days (Weeks 13-24)
Description: Monthly migraine days are summarized in 28-day intervals, and averaged across Weeks 13-24.
Time Frame: Week 13-24
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: Migraine Days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
Migraine Days | -9.0 (6.72) | -8.3 (7.03) | -6.4 (7.16)

14. Secondary Outcome: Change From Baseline in Monthly Headache Days (Weeks 1-12)
Description: Monthly headache days are summarized in 28-day intervals, and averaged across Weeks 1-12.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: Headache Days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
Headache Days | -8.8 (6.10) | -8.2 (5.78) | -6.4 (5.99)

15. Secondary Outcome: Time to First Migraine After Dosing
Description: The time to first migraine after dosing based upon the migraine data entered into the eDiary
Time Frame: 32 weeks
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
days | 4.0 [1.0 to 11.0] | 4.0 [1.0 to 9.0] | 2.0 [1.0 to 5.0]

16. Secondary Outcome: Change From Baseline to Week 12 in Percentage of Migraines With Use of Acute Medication
Description: The percentage of migraines with acute medication usage. Participants with no migraine will be included with a rate of zero.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: percentage of acute medication migraines
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
percentage of acute medication migraines | -14.10 (28.86) | -9.79 (26.78) | -2.82 (20.94)

17. Secondary Outcome: Change From Baseline to Week 12 in Percentage of Headaches With Use of Acute Medication
Description: The percentage of headaches with acute medication usage. Participants with no headaches will be included with a rate of zero.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: percentage of acute medication headaches
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
percentage of acute medication headaches | -7.46 (23.32) | -3.08 (21.31) | -0.16 (19.12)

18. Secondary Outcome: Percent Change in Frequency of Migraine Days - Week 1-12
Description: The percent change in frequency of migraine days from Weeks 1-12 was calculated as the number of migraine days within 4-week intervals that were then averaged up to Week 12. The difference of this estimate from baseline was calculated as the change from baseline in the frequency of migraine days over Weeks 1-12.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: percent change of migraine days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
percent change of migraine days | -53.5 (35.46) | -48.6 (36.60) | -34.5 (38.17)

19. Secondary Outcome: Percent Change in Frequency of Headache Days - Week 1-12
Description: The percent change in frequency of headache days from Weeks 1-12 was calculated as the number of headache days within 4-week intervals that were then averaged up to Week 12. The difference of this estimate from baseline was calculated as the change from baseline in the frequency of headache days over Weeks 1-12.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: percent change of headache days
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
percent change of headache days | -44.1 (30.59) | -41.2 (29.20) | -31.4 (28.62)

20. Secondary Outcome: Change From Baseline in Percentage of Severe Migraines
Description: The change from baseline in percentage of migraines that are classified as severe over Weeks 1-12.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: percentage of migraines scored "severe"
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
percentage of migraines scored "severe" | -18.17 (27.90) | -16.39 (26.17) | -10.82 (25.73)

21. Secondary Outcome: Change From Baseline in Percentage of Severe Headache
Description: The change from baseline in percentage of headaches that are classified as severe over Weeks 1-12.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: percentage of headaches scored "severe"
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
percentage of headaches scored "severe" | -14.00 (22.50) | -14.01 (20.95) | -9.12 (22.12)

22. Secondary Outcome: Change From Baseline in Monthly Migraine Hours, Weeks 1-12
Description: Migraine hours are the sum of migraines within 4 week intervals, and the average 4 week duration within 12 weeks.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: migraine hours
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
migraine hours | -80.9 (89.17) | -75.2 (90.40) | -52.8 (101.82)

23. Secondary Outcome: Change From Baseline in Monthly Headache Hours, Weeks 1-12
Description: Headache hours are the sum of the duration of headaches within 4 week intervals, and the average 4 week duration within 12 week intervals.
Time Frame: Week 1-12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: headache hours
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
headache hours | -82.5 (88.85) | -74.6 (84.57) | -54.8 (97.15)

24. Secondary Outcome: Duration of Migraine-Free Intervals
Description: The number of participants with migraine-free intervals starting within the first 2 weeks of treatment. The longest migraine free interval for each participant is recorded.
Time Frame: 32 weeks
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 350 | 356 | 366
Participants
  <= 7 days | 132 | 146 | 226
  8-14 days | 86 | 95 | 75
  15-21 days | 38 | 42 | 23
  >21 days | 94 | 73 | 42

25. Secondary Outcome: Change From Baseline of Short Form Health Survey (SF-36 v 2.0) Scale Scores
Description: The SF-36 is a health survey containing 36 questions consisting of eight scaled scores to measure quality of life over the past 4 weeks. All scales are on a range of 0 to 100, with 0 being the worst and 100 being the best. Scales are reported separately. Increases from baseline indicate improvement.
Time Frame: Baseline to Week 12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 338 | 343 | 343
score on a scale
  Physical Functioning | 3.3 (6.22) | 2.6 (5.98) | 1.5 (6.88)
  Role Physical | 6.0 (8.46) | 4.6 (8.53) | 3.6 (8.08)
  Bodily Pain | 6.2 (8.71) | 5.1 (9.12) | 4.0 (8.55)
  General Health | 3.5 (7.45) | 2.3 (6.89) | 0.7 (7.53)
  Vitality | 4.5 (9.02) | 4.2 (8.84) | 2.3 (8.23)

26. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 12
Description: The PGIC includes a single question concerning the participant's impression of the change in their disease status since the start of the study. Seven responses are possible: Very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse.
Time Frame: Week 12
Population: Full Analysis Population - all randomized participants who received investigational product or placebo. The Week 12 scores only include participants who completed the Week 12 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 337 | 344 | 343
Participants
  Very Much Improved | 73 | 54 | 38
  Much Improved | 142 | 126 | 92
  Minimally Improved | 68 | 82 | 85
  No Change | 51 | 69 | 111
  Minimally Worse | 3 | 10 | 16
  Much Worse | 0 | 2 | 1
  Very Much Worse | 0 | 1 | 0

27. Secondary Outcome: Health Related Quality of Life (EQ-5D-5L) at Week 12
Description: The EQ-5D-5L is a descriptive system of health-related quality of life states consisting of 5 dimensions/questions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses. The responses record five levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension.
Time Frame: Week 12
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
Number analyzed (Participants) | 338 | 344 | 343
Participants
  Mobility: No problems | 289 | 289 | 298
  Mobility: Slight Problems | 41 | 41 | 37
  Mobility: Moderate Problems | 8 | 13 | 6
  Mobility: Severe Problems | 0 | 1 | 2
  Mobility: Extreme Problems | 0 | 0 | 0
  Self-care: No problems | 320 | 337 | 331
  Self-care: Slight Problems | 13 | 6 | 7
  Self-care: Moderate Problems | 5 | 1 | 4
  Self-care: Severe Problems | 0 | 0 | 1
  Self-care: Extreme Problems | 0 | 0 | 0
  Usual Activities: No problems | 227 | 233 | 241
  Usual Activities: Slight Problems | 79 | 78 | 71
  Usual Activities: Moderate Problems | 27 | 28 | 26
  Usual Activities: Severe Problems | 5 | 5 | 4
  Usual Activities: Extreme Problems | 0 | 0 | 1
  Pain/Discomfort: No problems | 122 | 121 | 130
  Pain/Discomfort: Slight Problems | 140 | 127 | 120
  Pain/Discomfort: Moderate Problems | 56 | 78 | 75
  Pain/Discomfort: Severe Problems | 18 | 14 | 16
  Pain/Discomfort: Extreme Problems | 2 | 4 | 2
  Anxiety/Depression: No problems | 220 | 227 | 219
  Anxiety/Depression: Slight Problems | 91 | 87 | 91
  Anxiety/Depression: Moderate Problems | 23 | 25 | 27
  Anxiety/Depression: Severe Problems | 4 | 5 | 5
  Anxiety/Depression: Extreme Problems | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline to Week 32 (end of study)
Arm/Group | 300 mg ALD403 | 100 mg ALD403 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/350 | 0/356 | 0/366
Serious Adverse Events (participants affected / at risk) | 4/350 | 3/356 | 3/366
Other Adverse Events (participants affected / at risk) | 52/350 | 34/356 | 42/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg ALD403 (N=350) | 100 mg ALD403 (N=356) | Placebo (N=366)
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Migraine With Aura (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Depression Suicidal (Psychiatric disorders) | 0 | 1 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg ALD403 (N=350) | 100 mg ALD403 (N=356) | Placebo (N=366)
Nasopharyngitis (Infections and infestations) | 33 | 19 | 22
Upper respiratory tract infection (Infections and infestations) | 19 | 15 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT02974153/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT02974153/SAP_001.pdf